CLINICAL TRIAL: NCT03520153
Title: Characterization of Diabetes Mellitus in Fibrous Dysplasia/McCune-Albright Syndrome
Status: Withdrawn | Type: Observational
Why Stopped: The principal investigator is leaving Yale University and will not be continuing the work at her new institution.
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Other Study IDs: 2000022658
Record Dates: First submitted 2018-04-26; First posted 2018-05-09 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-07

CONDITIONS: McCune-Albright Syndrome; Fibrous Dysplasia; Intraductal Papillary Mucinous Neoplasm; Diabetes Mellitus
MeSH Terms: conditions — Fibrous Dysplasia, Polyostotic; Fibrous Dysplasia of Bone; Diabetes Mellitus | interventions — Glucose Tolerance Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- FD/MAS with diabetes mellitus: Fibrous Dysplasia/McCune-Albright Syndrome with diabetes mellitus.
  Participants will receive the following interventions: Hyperinsulinemic Euglycemic Clamp and 2H20; Hyperglycemic Clamp; and Oral Glucose Tolerance Test.
  Interventions: Procedure: Hyperinsulinemic Euglycemic Clamp and 2H20; Procedure: Hyperglycemic Clamp; Diagnostic Test: Oral Glucose Tolerance Test
- FD/MAS without diabetes mellitus: Fibrous Dysplasia/McCune-Albright Syndrome without diabetes mellitus.
  Participants will receive the following interventions: Hyperinsulinemic Euglycemic Clamp and 2H20; Hyperglycemic Clamp; and Oral Glucose Tolerance Test.
  Interventions: Procedure: Hyperinsulinemic Euglycemic Clamp and 2H20; Procedure: Hyperglycemic Clamp; Diagnostic Test: Oral Glucose Tolerance Test
- FD/MAS without diabetes and without IPMN: Fibrous Dysplasia/McCune-Albright Syndrome without diabetes mellitus and without intraductal papillary mucinous neoplasms.
  Participants will receive the following interventions: Hyperinsulinemic Euglycemic Clamp and 2H20; Hyperglycemic Clamp; and Oral Glucose Tolerance Test.
  Interventions: Procedure: Hyperinsulinemic Euglycemic Clamp and 2H20; Procedure: Hyperglycemic Clamp; Diagnostic Test: Oral Glucose Tolerance Test
- FD/MAS without diabetes and with IPMN: Fibrous Dysplasia/McCune-Albright Syndrome without diabetes mellitus and with intraductal papillary mucinous neoplasms.
  Participants will receive the following interventions: Hyperinsulinemic Euglycemic Clamp and 2H20; Hyperglycemic Clamp; and Oral Glucose Tolerance Test.
  Interventions: Procedure: Hyperinsulinemic Euglycemic Clamp and 2H20; Procedure: Hyperglycemic Clamp; Diagnostic Test: Oral Glucose Tolerance Test
- Healthy Controls: Participants will receive the following interventions: Hyperinsulinemic Euglycemic Clamp and 2H20; Hyperglycemic Clamp; and Oral Glucose Tolerance Test.
  Interventions: Procedure: Hyperinsulinemic Euglycemic Clamp and 2H20; Procedure: Hyperglycemic Clamp; Diagnostic Test: Oral Glucose Tolerance Test

INTERVENTIONS:
Procedure: Hyperinsulinemic Euglycemic Clamp and 2H20 — Test is used to assess insulin effects on hepatic glucose production.
Procedure: Hyperglycemic Clamp — Test of beta-cell function and insulin secretion. Involves increasing and maintaining blood glucose concentration with IV variable infusion of dextrose.
Diagnostic Test: Oral Glucose Tolerance Test — The oral glucose tolerance test (OGTT) measures the body's ability to use a type of sugar, called glucose, that is the body's main source of energy. An OGTT can be used to diagnose prediabetes and diabetes.

SUMMARY:
The investigators' objective is to understand the pathogenesis of diabetes mellitus in Fibrous dysplasia/McCune-Albright syndrome (FD/MAS) by: 1) establishing the contributions of insulin resistance versus impaired insulin secretion, 2) investigating presence of excess glucagon signaling by measuring gluconeogenesis and glycogenolysis, and 3) investigating a potential interaction between diabetes and intraductal papillary mucinous neoplasms (IPMNs).

DETAILED DESCRIPTION:
Specific project aims include:

Aim 1: Determine insulin secretion and sensitivity in subjects with MAS-associated diabetes.

Aim 2: Measure gluconeogenesis and glycogenolysis in MAS-associated diabetes to investigate a potential role for excess glucagon signaling.

Aim 3: Determine if IPMN development is associated with impairment of insulin secretion prior to development of overt diabetes.

The authors expect that this study will:

1. Establish the etiology of diabetes in FD/MAS
2. Increase understanding of the role of IPMNs in pathogenesis of diabetes
3. Provide critical insights into the pathogenesis of diabetes in FD/MAS

ELIGIBILITY:
Inclusion Criteria:

Fibrous dysplasia/McCune-Albright syndrome (FD/MAS) group:

* Must be diagnosed based on clinical grounds and/or mutation testing on bone and/or affected tissue

Control group:

* Must be at least 18 years old

Exclusion Criteria:

Fibrous dysplasia/McCune-Albright syndrome (FD/MAS) group:

* Unwilling to fully cooperate with the evaluation
* Unable to provide informed consent

Control group:

* History of diabetes, insulin resistance, pancreatic disease, pancreatic cysts or amylase/lipase abnormality
* Use of any type of oral diabetes medications and/or insulin
* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will include adult Fibrous dysplasia/McCune-Albright syndrome (FD/MAS) subjects (> 18 years-old) with diabetes, without diabetes, with and without intraductal papillary mucinous neoplasms (IPMNs). FD/MAS subjects, who are enrolled in the National Institutes of Health (NIH) Natural History Study and who have already been screened with an MRI of the abdomen or magnetic resonance cholangiopancreatography for pancreatic lesions, will be invited to participate in the current study based on an existing diagnosis of diabetes and/or IPMNs. In addition, seven adult healthy volunteers will be screened and recruited by the investigator from Yale Center for Clinical Investigation (YCCI) Recruitment Database.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-08-07 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Glucose tolerance status | Baseline
  An oral glucose tolerance test will be performed to assess glucose tolerance status to determine if subjects have pre-IGT, IGT or diabetes
Insulin sensitivity | Baseline
  This primary outcome will be obtained from the oral glucose tolerance test
Insulin secretion | Baseline
  This primary outcome will be obtained from the hyperglycemic clamp
Beta cell capacity | Baseline
  AIRmax stimulation test during the hyperglycemic clamp to ascertain the maximal acute insulin response (AIR) to arginine, which is a measure of functional beta cell capacity.
Hepatic glucose fluxes (gluconeogenesis and glycogenolysis) | At least 2 weeks post baseline testing
  Measurements from the Hyperinsulinemic Euglycemic Clamp/ 2H20 Study will be used to assess insulin effects on hepatic glucose production and glycerol kinetics isotopes and the deuterium enrichment at carbons 2 and 5 (C2 and C5) of plasma glucose providing information on glucose fluxes

SECONDARY OUTCOMES:
Islet cell antibodies (ICA), | Baseline
  Peripheral blood draw before the start of oral glucose tolerance test
Glutamic acid decarboxylase antibodies (GAD65) | Baseline
  Peripheral blood draw before the start of oral glucose tolerance test
Islet antigen-2 antibodies (IA-2A) | Baseline
  Peripheral blood draw before the start of oral glucose tolerance test
Zinc transporter 8 (ZnT8) | Baseline
  Peripheral blood draw before the start of oral glucose tolerance test
Fasting lipid panel | Baseline
  Peripheral blood draw before the start of oral glucose tolerance test
Fasting incretins | Baseline
  Peripheral blood draw before the start of oral glucose tolerance test
Prandial incretins | Baseline
  Peripheral blood draw at the end of the oral glucose tolerance test
Free fatty acids | Baseline
  Peripheral blood draw before the start of oral glucose tolerance test
Growth hormone | Baseline
  Peripheral blood draw before the start of oral glucose tolerance test
Insulin-like growth factor-1 (IGF-1) | Baseline
  Peripheral blood draw before the start of oral glucose tolerance test
Renal function (BUN and creatinine) | Baseline
  Peripheral blood draw before the start of oral glucose tolerance test
Hemoglobin A1c | Baseline
  Peripheral blood draw before the start of oral glucose tolerance test
Urinalysis | Baseline
  Will be obtained at baseline before the start of oral glucose tolerance test to look for albuminuria
Glycerol | Baseline
  Peripheral blood draw before the start of oral glucose tolerance test
Leptin | Baseline
  Peripheral blood draw before the start of oral glucose tolerance test
Adiponectin | Baseline
  Peripheral blood draw before the start of oral glucose tolerance test
Liver function tests (AST and ALT) | Baseline
  Peripheral blood draw before the start of oral glucose tolerance test
C-reactive protein (CRP) | Baseline
  Peripheral blood draw before the start of oral glucose tolerance test
Interleukin 6 (IL-6) | Baseline
  Peripheral blood draw before the start of oral glucose tolerance test
Tumor necrosis factor alpha (TNF-alpha) | Baseline
  Peripheral blood draw before the start of oral glucose tolerance test

OTHER OUTCOMES:
Maturity-Onset Diabetes of Young (MODY) genetic testing | Baseline
  The test detects deletions in the HNF4A, GCK, HNF1A, HNF1B genes and mutations in the HNF4A, GCK, HNF1A, HNF1B and IPF1. Will be obtained at baseline before the start of oral glucose tolerance test only in those subjects with an existing diagnosis of diabetes mellitus.

CONTACTS AND LOCATIONS:
Overall Officials: Cemre Robinson, MD, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States